CLINICAL TRIAL: NCT02077244
Title: A Randomized Controlled Trial to Evaluate the Effect of Nurse Led Follow up After Being a Patient in the Intensive Care Unit.
Brief Title: Follow up After Intensive Care. The FUTstudy
Acronym: FUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kirsti Tøien, PhD post doctor fellow, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012/1715
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-05

CONDITIONS: Post Traumatic Stress Symptoms; Post ICU Patient
Keywords: patient; intensive care; follow up; post traumatic stress symptoms; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Those who give their written informed consent will fill out the Post Traumatic Stress Scale 10 Intensive care screen (PTSS 10-I) Patients with a score equal or above 25 (indicating suffering from PTS symptoms) will be randomized to intervention or control group. Randomization will be performed using the computer program WebCRFNTNU. Patients who score below 25 will be included in an observation group and receive questionnaires at the same time points as the intervention and control group.
  To be able to detect a difference of 10 between the groups as significant with 80% power and allow for 20% dropout, a total of 250 patients with PTS-10 score like or above 25 have to be included in the randomized part of the study. In the autum 2016 a new statistician in the procject recalculated the power and found the need for 134 randomized patients. The inclusion was then terminated.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Follow up talks (Experimental): Patients with a score like or above 25 on Post traumatic stress scale-10 Intensive Care Screen after discharge from the ICU. Nurse led follow up talks at the ward and one and two months later.
  Interventions: Behavioral: Follow up talks
- No talks (No Intervention): Patients with a score like or above 25 on Post traumatic stress scale-10 Intensive Care Screen after discharge from the ICU. Care as usual
- Observation group (No Intervention): Patients with a score below 25 on Post traumatic stress scale-10 Intensive Care Screen after discharge from the ICU. Care as usual.

INTERVENTIONS:
Behavioral: Follow up talks — Nurse led follow up talks at the ward and one and two months later.
  Arms: Follow up talks

SUMMARY:
To investigate the effect of nurse led follow up talks to prevent posttraumatic stress (PTS) symptoms and improve quality of life and sence of coherence after an intensive care unit (ICU) stay.

Secondly:

Investigate level of psychological distress, quality of life, hope and work participation in ICU patients after an ICU stay and factors associated with these outcomes.

DETAILED DESCRIPTION:
The ICU patient experiences total dependence on health care professionals and technical devices. Some patients report unpleasant memories such as pain, feeling helpless, or delusional experiences from the ICU stay and many report physical or mental symptoms after discharge from the ICU. Return to work rate after ICU treatment differs. Most ICU patients receive analgesics and sedatives to relieve pain and discomfort during the stay. Thus many patients have few memories from their time being critically ill. For patients with few memories from the ICU stay this represents an interruption in the patient's life history. Since personal identity is influenced by the stories we tell about ourselves, loss of memory from a period with critical illness might be experienced as a threat towards self-confidence and sense of coherence. Some patients with traumatic memories from the ICU develop PTS symptoms after discharge.

In order to help the earlier ICU patient to achieve a life with less physical and mental complaints, some ICUs have established a follow up program in outpatient clinics after discharge from hospital, but there is sparse evidence of the effectiveness of this intervention, and what type of follow up that best help the patients.

The primary aim of the study is to:

Investigate if a group of previous intensive care patients receiving nurse led follow up talks three times after discharge from the ICU have less post traumatic stress symptoms, pain, increased sense of coherence and, work participation and health related quality of life (HRQL) three, six and twelve months after discharge from the ICU compared to a control group receiving standard care.

Secondary aim:

Investigate level and predictors of anxiety, depression, PTS symptoms, hope, pain, HRQOL and work participation in intensive care patients ICU patients first year after discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an ICU stay like or above 24 hours who speak and understand Norwegian and who are conscious and cognitively oriented at the time of inclusion. Patients with a score of 25 or more on Post Traumatic Stress Scale 10 (PTSS-10) is randomized to intervention or control group. Patients with a score below 25 on PTSS-10 is included in an observation group.

Exclusion Criteria:

* severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress symptoms | 3, 6 and 12 months after baseline
  Baseline is measured when the patient has been discharged from the ICU to a ward. Change from baseline at 3, 6 and 12 months.

SECONDARY OUTCOMES:
Sense of coherence (Sense of coherence scale 13) | 3, 6 and 12 months after baseline
  Baseline is measured when the patient has been discharged from the ICU to a ward. Change from baseline at 3, 6 and 12 months.
Health related quality of life | 3, 6 and 12 months after baseline
  Baseline is measured when the patient has been discharged from the ICU to a ward. Change from baseline at 3, 6 and 12 months.
Pain (Brief pain inventory) | 3, 6 and 12 months after baseline
  Baseline is measured when the patient has been discharged from the ICU to a ward before leaving the hospital. Change from baseline at 3, 6 and 12 months.
Work participation | 3, 6 and 12 months after baseline
  Baseline is measured when the patient has been discharged from the ICU to a ward. Change from baseline at 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway